CLINICAL TRIAL: NCT05897021
Title: Expressive Writing to Reduce Depressive and Anxiety Symptoms Among Sexual Minority Veterans
Brief Title: Expressive Writing on Minority Stressors Among Sexual Minority Veterans
Acronym: EWMS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MHBC-008-22F; IK2CX002629 (NIH)
Record Dates: First submitted 2023-06-01; First posted 2023-06-09 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Depressive Symptoms; Anxiety
Keywords: Sexual Minorities; Veterans; Depressive Symptoms; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: In Phase I, all sexual minority Veterans will receive EWMS, which will be iteratively refined based on qualitative interviews at end of treatment, consultation with experts in sexual minority health (Dr. Livingston and SMEs, Drs. Sloan and Pachankis) and discussion amongst mentors (Drs. Marx, Livingston, and Iverson).
  In Phase II, sexual minority Veterans who are eligible (i.e., clinically significant depression and/or anxiety symptoms and a history of sexual minority stressor exposure that is reported by Veterans to be related to their distress) will be randomized to the EWMS condition or to the neutral control condition. Participants will complete the assigned intervention condition and will be assessed at baseline, post-treatment, and 3 month follow-up.
Who Masked: Outcomes Assessor
Masking Description: Outcome Assessors will be independent from the Study Team and will be blind to participants' treatment condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Expressive Writing on Minority Stressors (Experimental): The EWMS protocol will consist of 3 sessions delivered by a therapist (either in-person or remotely via telehealth platform) to sexual minority Veterans. The intervention will begin with an overview of the intervention, brief psychoeducation about expressive writing, and a review of the potential benefits of expressive writing. The initial session will also consist of psychoeducation on sexual minority stressors and common reactions to these stressors (i.e., universal stress reactions and minority-identity specific reactions) and how this relates to psychological outcomes, such as depression and anxiety, and high-risk behaviors, such as substance use and suicidal ideation. The initial session will be 60 minutes (introduction, psychoeducation, and first writing exercise) and the following two sessions (feedback, writing exercises, and check-ins) will take approximately 40 minutes.
  Interventions: Behavioral: Expressive Writing on Minority Stressors
- Neutral Writing (Placebo Comparator): To be comparable to EWMS, the control intervention will also be a 3-session individual intervention involving engaging in a writing exercise per session. For the control writing exercises, participants will be asked to write for 30 minutes about their daily activities since waking up that day based on Pennebaker's standard writing paradigm (Pennebaker & Beall, 1987). Individuals in the control condition will also be given information about the purpose of the writing exercises to be comparable to the psychoeducation information provided in EWMS. Similar to EWMS, the clinician will check in with the participant about the writing session, such as asking how the session went and how it felt to do the writing, following the 30 minutes of writing.
  Interventions: Behavioral: Neutral Writing

INTERVENTIONS:
Behavioral: Expressive Writing on Minority Stressors — The EWMS protocol will consist of 3 sessions delivered by a therapist (either in-person or remotely via telehealth platform) to sexual minority Veterans. The intervention will begin with an overview of the intervention, brief psychoeducation about expressive writing, and a review of the potential benefits of expressive writing. The initial session will also consist of psychoeducation on sexual minority stressors and common reactions to these stressors (i.e., universal stress reactions and minority-identity specific reactions) and how this relates to psychological outcomes, such as depression and anxiety, and high-risk behaviors, such as substance use and suicidal ideation. The initial session will be 60 minutes (introduction, psychoeducation, and first writing exercise) and the following two sessions (feedback, writing exercises, and check-ins) will take approximately 40 minutes.
  Arms: Expressive Writing on Minority Stressors
Behavioral: Neutral Writing — To be comparable to EWMS, the control intervention will also be a 3-session individual intervention involving engaging in a writing exercise per session. For the control writing exercises, participants will be asked to write for 30 minutes about their daily activities since waking up that day based on Pennebaker's standard writing paradigm (Pennebaker & Beall, 1987). Individuals in the control condition will also be given information about the purpose of the writing exercises to be comparable to the psychoeducation information provided in EWMS. Similar to EWMS, the clinician will check in with the participant about the writing session, such as asking how the session went and how it felt to do the writing, following the 30 minutes of writing.
  Arms: Neutral Writing

SUMMARY:
Sexual minority stressors (e.g., sexual minority identity-based discrimination) contribute to greater risk for and severity of depression, anxiety, substance use disorders and suicide among sexual minority Veterans. However, no brief, scalable, one-on-one interventions targeting sexual minority stressor-related distress are available in Veterans Affairs (VA) for sexual minority Veterans. The proposed research will examine the feasibility, acceptability, and preliminary effectiveness of a brief, 3-session expressive writing intervention to target distress related to sexual minority stressor exposure among sexual minority Veterans. The results of this work will advance knowledge about a promising brief and easy to implement intervention focused on reducing depressive and anxiety symptoms among sexual minority Veterans. This proposal aligns with VA's and CSR&D's commitment to providing equitable services to sexual minority Veterans and the aim of reducing health disparities among underserved Veteran groups.

DETAILED DESCRIPTION:
Sexual minority Veterans (e.g., gay, lesbian, bisexual) are one of the highest risk populations for psychiatric disorders due in part to the experience of discrimination and stigma-based stressors (sexual minority stressors). These stressors and the associated stress responses contribute to greater severity of depression and anxiety, which confer risk for negative health outcomes (hazardous substance use and suicide). However, very few interventions target distress related to sexual minority stressors, and even fewer have been tested in Veteran Health Administration (VHA). Brief, easy to implement interventions that target distress related to sexual minority stressors are needed to address the unique mental health concerns of this high risk community of Veterans. Expressive writing is a brief, well-developed paradigm that involves writing about thoughts and emotions related to a stressful experience for at least 15 minutes, 3-5 times based on a structured writing prompt. Over 30 years of research supports expressive writing's effectiveness in reducing stress, depression, and anxiety related to a stressor. Expressive writing on a minority stressor (EWMS) has been shown to reduce depression and anxiety among sexual minority non-Veterans but has never been tested among sexual minority Veterans. The aim of the proposed study is to examine the feasibility, acceptability, and preliminary effectiveness of EWMS, a promising intervention for sexual minority Veterans. Based on consultation with experts in expressive writing and sexual minority Veteran health, EWMS will be adapted for sexual minority Veterans and a VHA clinic setting. EWMS will be implemented as a 3 session, one-on-one intervention with a therapist. The proposed EWMS protocol will be iteratively refined in a case series (n = 10), and then tested in a pilot randomized control trial (RCT; n = 54) comparing EWMS to a neutral writing control condition. Aims of the pilot RCT are: 1) demonstrate feasibility and acceptability of study procedures and EWMS using quantitative and qualitative data; and 2) examine the preliminary effectiveness of EWMS relative to control in reducing depressive and anxiety symptom severity. The proposed research aims are in direct alignment with the applicant's short term and long term training goals. The proposed research and complimentary mentorship and training plans will enable the applicant to: 1) gain expertise in intervention adaptation and clinical trial research; 2) gain expertise in sexual minority health; 3) develop aptitude in implementation theory and processes to inform future implementation of the proposed intervention and other interventions; and 4) achieve career independence. The results of the pilot RCT along with the training and mentorship of this project will inform a Merit award submission comparing EWMS with an active control in a hybrid I implementation-effectiveness trial to test the efficacy of the intervention while collecting information on barriers and facilitators to implementation of the intervention. This proposed research, training, and mentorship plan will provide the applicant with the necessary skills and experience to transition into an independent clinical researcher in VA focused on the development, enhancement, and implementation of interventions for minority related stress among sexual minority Veterans. The research and training will take place at the National Center for Posttraumatic Stress Disorder at the VA Boston Healthcare System under the supportive, collaborative, and accomplished mentorship team, including Drs. Brian Marx (primary mentor), Katherine Iverson (co-mentor), and Nicholas Livingston (co-mentor). These mentors have unique, yet complimentary, areas of expertise and have an established and successful history working together and with the applicant. The research, mentorship, and training proposed will facilitate the applicant's transition into a successful and productive independent VA investigator conducting research that directly aligns with VA's priority to provide equitable, patient-centered services to Veterans.

ELIGIBILITY:
Inclusion Criteria:

Participants will be Veterans who:

* identify as a sexual minority (i.e., identify as gay, lesbian, bisexual, pansexual, queer, or another identity other than heterosexual)
* endorse clinically significant depressive or anxiety symptoms (score above 10 on the PHQ-9 or GAD-7)
* report a history of sexuality-based minority stressor exposure that is contributing to distress on phone screening
* be stable on psychotropic medication for at least 4 weeks if on a psychotropic medication

Exclusion Criteria:

The exclusion criteria for Veterans in this study are:

* clear and current suicidal plan and/or intent (assessed via the Columbia Suicide Severity Rating Scale)
* current presentation of unstable mania and/or psychosis (assessed via the Structured Interview for DSM-5)
* current substance use disorder, severe (assessed via the Structured Interview for DSM-5)
* significant cognitive impairment, including evidence of moderate or severe traumatic brain injury, determined by an inability to comprehend baseline screening questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the Expressive Writing on Minority Stressors (EWMS) intervention | This will be assessed through study completion at the end of Phase II of the Study (i.e., end of the 4th year)
  Level of feasibility will be assessed by comparable percentage of treatment completion as found in a previous efficacy trial of Expressive Writing on Minority Stressors in a non-Veteran sample (Pachankis et al., 2021). The percentage of treatment completion will be comparable to percentage of treatment completion reported in a previous efficacy trial of EWMS with young adults (89%) (Pachankis et al., 2021).
Patient satisfaction with the Expressive Writing on Minority Stressors (EWMS) intervention | Veterans will complete the Client Satisfaction Questionnaire at the post-treatment (3-4 weeks after beginning treatment) assessment
  Veterans who are assigned to the EWMS condition will report comparable levels of treatment satisfaction on the Client Satisfaction Questionnaire-8 (CSQ-8; Larsen et al., 1979) as other efficacy trials using expressive writing paradigms (Sloan et al., 2012).

SECONDARY OUTCOMES:
Depressive symptom severity on the Patient Health Questionnaire-9 (PHQ-9) | baseline, post-treatment (3-4 weeks after beginning treatment), and 3-month follow-up
  The PHQ is a 9-item self-report measure of depression symptoms, and includes an item assessing suicidal ideation. Administered at baseline, posttreatment, and follow-up.
  Repeated measures analysis of variance (ANOVA) models will be used to detect group mean differences in depression symptom severity at the 3-month follow-up. The investigators will treat time (baseline, post-treatment, 3-month follow-up) as the within variable and group (i.e., EWMS vs. neutral control) as the between variable, and include the interaction of time and condition in the model. If the interaction between time and condition is significant, the investigators will conduct post hoc analysis with a Bonferroni adjustment to compare group mean differences in depressive symptom severity.
Anxiety symptom severity based on the Generalized Anxiety Disorder-7 (GAD-7) | baseline, post-treatment (3-4 weeks after beginning treatment), and 3-month follow-up
  The GAD7 is a 7-item self-report measure of anxiety symptoms. Administered at baseline, posttreatment, and follow-up.
  Repeated measures analysis of variance (ANOVA) models will be used to detect group mean differences in anxiety symptom severity at the 3-month follow-up. The investigators will treat time (baseline, post-treatment, 3-month follow-up) as the within variable and group (i.e., EWMS vs. neutral control) as the between variable, and include the interaction of time and condition in the model. If the interaction between time and condition is significant, the investigators will conduct post hoc analysis with a Bonferroni adjustment to compare group mean differences in anxiety symptom severity.

CONTACTS AND LOCATIONS:
Overall Officials: Kelly L Harper, PhD, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (1):
- VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No